CLINICAL TRIAL: NCT06782464
Title: Ultrasound Guided Cryoneurolysis to Treat Shoulder Pain and Functional Problems Related to Upper Limb Spasticity
Brief Title: Upper Limb Nerve Cryoneurolysis is Non Inferior to the Usual Care and Has Therapeutic Add Value in Dealing with Shoulder Pain and Functional Problems Caused by Spasticity and Motor Impairment
Acronym: spastiCRYO-UL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre National de Rééducation Fonctionnelle et de Réadaptation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: spastiCRYO-UL
Record Dates: First submitted 2024-12-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Hemiplegia; Spasticity; Shoulder Spasticity; Shoulder Stiffness; Stroke; Multiple Sclerosis; Traumatic Brain Injury; Spinal Cord Injury
Keywords: cryoneurolysis; spasticity; pain; stroke; traumatic brain injury; spinal cord injury
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity; Stroke; Multiple Sclerosis; Brain Injuries, Traumatic; Spinal Cord Injuries; Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The upper limb clinical trial of the spastiCRYO research project is a multinational interventional randomized controlled trial. As stated previously, it compares the clinical effectiveness of an interventional session consisting in ultrasound guided peripheral pectoral lateral and thoracodorsal nerves cryoneurolysis plus an upper limb rehabilitation programme with the standard care, which is an interventional session consisting in BoNT-A intramuscular injection in pectoralis major, subscapularis and teres major muscles, plus an upper limb rehabilitation program, for the treatment of shoulder pain and functional problems caused by spasticity of the upper limb.
  Setting The trial is conducted in two Rehabilitation Hospitals in different countries (multicentric): In Portugal and Luxembourg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intramuscular injection of onabotulinumtoxinA (Active Comparator): Participants allocated to this group have intramuscular injections, guided by ultrasound and electrical neurostimulation, of BoNT-A (ona botulinum toxin A) to the pectoralis major (75 UI), subscapularis (75 UI) and teres major (50 UI), dilution 100UI/ml. These muscles selection and doses are chosen according to a literature review incriminating these 3 muscles as the responsible for a common spastic pattern of shoulder adduction and internal rotation and contributing to the shoulder pain.
  Interventions: Procedure: Treatment
- Ultrasound-guided Cryoneurolysis with Metrum Cryo-painless S device (Experimental): The cryoneurolysis intervention is performed by a trained and experienced physician. Ultrasound guided cryoneurolysis to the lateral pectoral nerve and to the thoracodorsal nerve is the intervention in this group. The 3 parts of the pectoral major muscle (clavicular, sternal and costal) innervated by different branches of the lateral pectoral nerve might be targeted as needed80.
  The cryoneurolysis device being used is the "Cryo-S Painless" produced by Metrum, a manufacturer based in Poland. The cryoprobes have a caliber of 1.3 mm. These devices hold medical certification (Conformité Européenne CE) for cryoanalgesia within the European Union.
  Technical and certification files are provided to the Regulatory agencies in Luxembourg.
  (https://www.metrum.com.pl/produkty/cryo-s-painless-2/?lang=en ). Several precautions steps are taken to prevent the incidence of adverse effects.
  Interventions: Procedure: Treatment

INTERVENTIONS:
Procedure: Treatment — Treatment

SUMMARY:
This trial is part of the spastiCRYO clinical research project. The primary objective of this clinical trial is to test the hypothesis: "Upper limb nerve cryoneurolysis is non inferior to the usual care and has therapeutic add value in dealing with shoulder pain and functional problems caused by spasticity and motor impairment".

It is a non-inferiority study on the referred topic, comparing the therapeutic effect (improvement in function and pain) of cryoneurolysis of selected nerves (lateral pectoral nerve and thoracodorsal nerve) with the usual care: intramuscular botulinum neurotoxin type A (BoNT-A) injection of pectoralis major, teres major and subscapularis muscles. The hypothesis is that cryoneurolysis is not inferior to the usual care in terms of magnitude of the therapeutic effect and might have a therapeutic add-value in terms of duration of that effect.

Two secondary hypotheses are firstly, that cryoneurolysis is a safe procedure that can be deployed in a rehabilitation hospital setting with minimum requirements to perform mini-invasive procedures and secondly that selecting patients who might benefit from this treatment is straightforward.

To test these hypotheses, the research team will gather, analyse and compare outcome measures data from the endpoints which are the changes along the trial duration in shoulder pain, upper limb function, involved muscles spasticity, shoulder range of motion (abduction and external rotation) level of impairment, and follow-up of potential adverse effects in two independent and equivalent groups of participants who have shoulder pain and functional limitations caused by spasticity and are in a stable phase of their condition. Participants in one group (cryoneurolysis arm) have one session of selected nerves ultrasound and neurostimulation guided cryoneurolysis and participants in the other group (BoNT-A arm) have one session of ultrasound and neurostimulation guided injection of BoNT-A in the pectoralis major, teres major and subscapularis.

The participants of the two groups follow an upper limb analogous rehabilitation program for 24 weeks after each intervention. Longitudinal follow-up in the trial will take 24 weeks. In a real-world scenario, within 24 weeks the effect of Bont-A intramuscular injection has already waned, and the procedure should be repeated.

Secondary objectives are to compare changes in upper limb sensory function and electroneuromyographic parameters with the intention to understand the cryoneurolysis mechanism of action and the reversibility of this mini-invasive intervention. Changes in quality-of-life dimension of participants is a secondary endpoint as well.

DETAILED DESCRIPTION:
Hypothesis and state of the art Spasticity is a common clinical feature in several central nervous system conditions (stroke, traumatic brain injury, spinal cord injury, multiple sclerosis cerebral palsy, etc.). Strictly, spasticity refers to the increased excitability of the phasic and tonic muscular stretch reflexes in the absence of volitional activity observed in patients with upper motor neuron lesion.

Gracies has eloquently explained that spasticity is one of the presentations of the pathological stretch-sensitive muscle overactivity in spastic paresis, the other two being spastic dystonia and muscle cocontraction. The muscle overactivity is a neurophysiological consequence of the motor command disruption and sensorimotor privation which, associated with muscle hypo-mobilization in short position is also responsible for the spastic myopathy . Nevertheless, in the literature, experts use interchangeably these concepts and spasticity is often employed as an umbrella term, a synonym of all the positive signs of the corticospinal (pyramidal) pathway disorder, referring to a broad spectrum of clinical manifestations as disorganization of motor volitional command, loss of motor selectivity, muscle overactivity with co-contractions, muscular synkinesis, aberrant synergic patterns, increased muscular tone, abnormal postures, clonus, deep tendon hyperreflexia, spasms and spastic dystonia.

Spasticity is often associated with sensory impairment. Long lasting spasticity left untreated leads to irreversible anatomical structural changes, including muscular tendon shortenings and imbalances, joint stiffness, or other musculoskeletal deformities as well as pain. For instance, in stroke survivors (2017: 9,53 million persons in EU) spastic paralysis and associated functional loss, along with cognition limitations are the most dramatic consequences that these persons, their caregivers and relatives must deal with. The number of people living with stroke is estimated to increase by 27% between 2017 and 2047 in the European Union, mainly because of population ageing and improved survival rates.

Spastic paresis and muscle hypertonia of the limbs caused by spasticity, expresses in different rigid postures, which, added to sensory impairment and motor control loss, is a source of dysfunction, pain and discomfort, leading to trophic deterioration, skin lesions and disrupted body image with negative impact in self-esteem. In these cases, it can even interfere with providing care for basic daily live activities (transfers, being dressed, hygienic care), and preclude fully social participation of persons having spasticity.

Quantifying the impact of spasticity at the organ level is a well-known issue and controversy still exists in non-instrumental measurements of spasticity and its treatment efficacy. Different scales are widely used with diverse intra and inter examiner variability. The challenge is even greater when there are several joints involved and a composite metric is needed. When evaluating the effects of a specific spasticity treatment, it is pertinent to consider the patients and therapeutic team's treatment goals. Likewise, the changes the treatment strategy might provoke in other dimensions as pain, trophic changes, social participation, self-esteem, caregiver burden, self-care, autonomy, and quality of life should be take into account.

Nowadays, there are several therapeutic interventions to manage functional and structural problems caused by spasticity. These options are usually applied in sequential combined protocols to achieve a balanced outcome between negative and positive functional outputs of a spastic limb. In the framework of the therapeutic escalation, the reversibility of the treatment must be considered. Invasive procedures that act directly or indirectly on the uninhibited muscle stretch reflex loop and are reversible to some degree include: (1) minimally invasive procedures such as intramuscular BoNT-A or chemical peripheral nerve denervation (chemodenervation) with alcohol and phenol, percutaneous tenotomies and (2) more invasive procedures such as neurosurgery (peripheral nerve neurotomy and neurectomy, selective dorsal rhizotomy, intrathecal baclofen pump implantation, and neuromodulation.

Other major invasive and irreversible procedures such as neuro-orthopaedic surgery (tendon transfers, soft tissue lengthening, correction of secondary skeletal deformities, and arthrodesis) may also be performed. Finally, non-invasive interventions exist such as physiotherapy, plaster casts, orthoses, functional electrical stimulation, neuroplasticity interventions, and pharmacological agents .

Most of those therapeutic options are costly in term of health resources (human, financial, operating theatre workflows, expensive pharmacological agents, risk exposure, hospital backlogs), not widely available and, should be addressed in an era of hospital staff shortages, supply chain bottlenecks and strained delivery of care.

In the therapeutical decision-making discussion, weighing the contribution to the active and passive loss of mobility, between the dynamic overactivity of the muscle versus the passive elements is crucial. This can be accomplished by a diagnostic nerve block (DNB). This intervention will knock-off temporarily the uninhibited myotatic stretch reflex, therefore, while the block lasts, the resulting resistance to movement is related to the altered passive viscoelastic properties of the muscle-fascia-tendon unit, and/or to the joint. Therefore, diagnostic motor block rules out structural and rheologic causes of stiffness. and at the same time it can simulate the result of a spasticity therapeutic intervention that targets muscle overactivity.

In a general population of stroke survivors, the prevalence of hemiplegic shoulder pain is approximately 22-23% and in a rehabilitation setting it is 54-55%, a majority of patients present moderate to severe pain and it correlates with reduction in quality of life . The etiology of post stroke hemiplegic shoulder pain is often not clear but it seems that spasticity of muscles controlling the shoulder plays an important role. Pectoralis major, teres major and subscapularis muscles are targets for BoNT-A injection as a treatment for hemiplegic shoulder pain.

Cryoneurolysis (also named cryoablation, cryoneurotomy, cryodenervation) is a biophysical controlled lesion of a peripheral nerve, provoked by focused cold generated by a specific medical device. The lowering of temperature between -30 to -40, is provoked by a cryoprobe creating an ice ball, from surrounding tissular water molecules, around the nerve in a specific location. The procedure is guided by ultrasound, and the cryoprobe can also make sensory and/or motor stimulation to finetune the selection of the targeted nerve.

This technology is indicated in peripheral nerves to create a long lasting locoregional anaesthesia in defined painful conditions. It creates a controlled damage by inducing ischemia in the nerve, leading to an axonotmesis leaving intact the perineurium and epineurium (2nd degree nerve lesion according to Sunderland) and therefore, allowing for a reparative process to undergo without a random proliferation of fibrotic scar and avoiding the neuroma formation. In interventional pain settings, a cryoneurolysis therapeutic session lasts about 30-45 minutes/patient and can be performed in an outpatient clinic.

There are some published preliminary applications of cryoneurolysis in spasticity in humans but still many unanswered questions persist, such as treatment efficacy and tolerance, defining the profile of cryoneurolysis indications and patient selection criteria in spasticity, establishing ideal biophysical parameters (number, duration of freezing cycles, ice ball size and distance from the targeted nerve), interest in targeting mixed peripheral nerves (sensory, motor, vegetative), risk exposure, etc, claiming further clinical investigation. As in interventional pain treatment, cryoneurolysis therapeutic effects in spasticity may wane, at an unknown rate, and it might be needed to repeat the procedure.

In a recent paper analysing adverse effects of cryoneurolysis in the treatment of spasticity in 113 patients (277 nerves), Winston et al state that cryoneurolysis has the potential to be a safe method of treating spasticity. Nevertheless in 7 out of 99 cryoneurolysed mixed motor/sensory nerves, patients developed dysesthesia that lasted a maximum of 3 months. Considering these findings, the investigators use exclusively motor nerves or motor nerve branches on our clinical trial protocol.

The American Academy of Physical Medicine & Rehabilitation (AAPM&R) recently published a consensus guidance on spasticity assessment and management, authored by Monica Verduzco-Gutierrez, M.D. et al. This paper eloquently summarizes the current state of the art in spasticity assessment and treatment. Notably, the authors mention cryoneurolysis as a potentially safe treatment for spasticity, though they emphasize that further studies are needed.

Our hypothesis is that ultrasound guided peripheral nerve cryoneurolysis, as a minimal invasive technique acting at the pathologically uninhibited myotatic loop, can be integrated in the therapeutic protocols to treat the shoulder functional limitations and pain caused by spasticity and that cryoneurolysis is not inferior in terms of therapeutic value and is safe and the therapeutic effects might last longer when compared to a standard of care in this condition (BoNT-A intramuscular injection).Risks/Benefits trade-off.

Cryoneurolysis of peripheral nerves offers several advantages for treating spasticity when compared to other therapeutic options. Unlike neurotomy-a surgical procedure-ultrasound-guided cryoneurolysis can be performed in an outpatient setting. This frees up operating theatre availability and reduces the need for specialized staff.

The research team has identified some distinct advantages of cryoneurolysis over intramuscular BoNT-A injections. First, cryoneurolysis has an immediate therapeutic effect and tends to last longer. Moreover, for complex spastic conditions, a systematic, step-by-step approach can be adopted. This involves sequencing cryoneurolysis procedures spaced about a week apart. Such a protocol lets patients witness the outcomes of one cryoneurolysis treatment, undergo further functional evaluation in real-world conditions or a movement laboratory, and if necessary, receive another treatment shortly thereafter to optimize results. This flexibility contrasts with BoNT-A injections, which require a minimum of a three-month interval between sessions. And finally, cryoneurolysis per se is a biophysical phenomenon not implying administration of drugs, without the risks of allergic reactions or antibody formation.

Compared to neurolysis using alcohol and phenol for spasticity treatment, cryoneurolysis offers a distinct advantage as it doesn't cause destruction or induce necrosis in neighbouring tissues such as fascia, muscles, and blood vessels. Moreover, phenol can lead to allergic reactions, neuroma formation, and exhibits caustic properties that can harm tissues.

Like all minimally invasive procedures, cryoneurolysis comes with inherent risks and potential side effects. However, when all safety protocols are diligently followed, these risks are substantially reduced. It's imperative that patients with certain conditions, including cryoglobulinemia, paroxysmal cold haemoglobinuria, cold urticaria, Raynaud's disease, or those with open and/or infected skin wounds, abstain from this treatment. Winston et al75 have highlighted potential complications from cryoneurolysis such as skin infections, bruising, swelling, and dysesthesia.

Dysesthesia, which persists for 4-6 weeks, is exclusively reported in approximately 7% of mixed nerves subjected to cryoneurolysis75. This sensation may arise from cold-induced neuropraxia, particularly impacting the sensory components of the treated nerves exposed to temperatures ranging from 0 to -20°C at the periphery of the ice ball. As a result, patients undergoing cryoneurolysis on mixed nerves require careful monitoring. Tailored treatments, such as neuropathic pain oral medications or ultrasound-guided peripheral nerve blocks with long-acting anaesthetics and corticosteroids, should be made available to them.

Condition or disease Post stroke, anoxic or traumatic brain injury, shoulder pain and functional problems caused and related to upper limb spasticity.

Principal Investigator

The Principal Investigator for Luxembourg is José Pereira M.D., while for Portugal, it's Dr. Simao Serrano M.D.

Institutions In Luxembourg, the spastiCRYO research project, which includes the upper limb clinical trial, is conducted at the Rehazenter. spastiCRYO is one of the ongoing clinical research projects within the RehaLAB, the Rehazenter Clinical Research Unit. Dr. Frederick Dierick, PhD, oversees research activities at RehaLAB in, while Céline Schreiber, Ing., manages the dataset and analysis.

In Portugal, the research team led by Simao Serrano, M.D., conducts the trial at the National Rehabilitation Center in Coimbra. Both institutions operate within the public economic sector.

At both institutions, the infrastructure and staff competencies, including nursing and adherence to standard hygiene, logistics, and safety protocols, are well-suited for all interventions in this trial.

Funding This clinical trial is incorporated into the participants' care plan and falls under the umbrella of the spastiCRYO research project.

In Luxembourg, this project receives financial backing from the Health Ministry, which funds 0,3 to 0.5 full-time equivalent during 4 years of the Principal Investigator, Dr. José Pereira.

Metrum, the industry partner for this trial, has generously provided the Metrum Cryo Painless device on loan and provides staff training and equipment maintenance at no cost for the trial's duration.

Study Design

Study type The upper limb clinical trial of the spastiCRYO research project is a multinational interventional randomized controlled trial. As stated previously, it compares the clinical effectiveness of an interventional session consisting in ultrasound guided peripheral pectoral lateral and thoracodorsal nerves cryoneurolysis plus an upper limb rehabilitation programme with the standard care, which is an interventional session consisting in BoNT-A intramuscular injection in pectoralis major, subscapularis and teres major muscles, plus an upper limb rehabilitation program, for the treatment of shoulder pain and functional problems caused by spasticity of the upper limb.

Setting The trial is conducted in two Rehabilitation Hospitals in different countries (multicentric): in the Centre National de Rééducation et de Réadaptation Fonctionnelle (Rehazenter) in Luxembourg and in the Centro de Medicina de Reabilitação da Região Centro Rovisco Pais (Centro de Reabilitação Rovisco Pais) in Portugal.

The privacy procedures and data storage respect the General Data Protection Regulation.

Enrolment Potential participants are identified through the routine clinical practices of physicians and therapeutic team members at the two rehabilitation hospitals involved in the study. Furthermore, referrals from other hospitals guide prospective participants to the screening assessment consultation for the clinical trial.

All potential candidates who choose not to participate in the clinical trial, as well as those who decide to withdraw after enrolment, will be provided with the standard of care for their respective health conditions.

Screening assessment consultation At their initial consultation, potential participants meet with the trial physician alongside a trusted individual they've designated beforehand, such as a family member or friend. This trusted individual is present throughout the visit to offer support and insight. The trial physician assesses eligibility criteria; if a subject meets any exclusion criteria, they are informed of the reason for their ineligibility, concluding their involvement in the trial.

Eligible participants receive detailed information about the trial's hypothesis, design (including the cryoneurolysis and BoNT-A arms and randomization process), objectives, setting, potential side effects, and risks. They are reassured that they have the freedom to withdraw from the trial whenever they wish. Furthermore, their decision to participate, withdraw, or drop out will not influence their standard care or treatment in any way. The privacy and data protection measures are also explained.

They are also informed that during the six-month trial, participants who do not respond to either intervention may withdraw from the study and will be offered an alternative treatment protocol. This could include changing the intervention or implementing other therapeutic options.

During this session, the physician gathers demographic and clinical data from the eligible participants. They are then introduced to the informed consent form. After this, both the participant and their designated trusted individual are given a reflection period and are presented with a written overview of the trial. If necessary, they can arrange a follow-up consultation with the physician to address any further questions. Only after reading, understanding, and signing the informed consent will participants advance to the trial's baseline evaluation.

Endpoints and Outcome Measures

The primary endpoint that this clinical trial aims to ascertain is the:

1. Improvement in shoulder external rotation passive range of motion The secondary endpoints to be ascertain are.
2. Changes in

i. Shoulder passive/active range of motion in Abduction ii. Muscle tone for shoulder internal rotators and adductors. iii. Pain (nociceptive and neuropathic) iv. Prehension / grasping / grip v. Quality of life c. Electromyographic changes in cryoneurolysed nerve(s)/corresponding muscles d. The degree of attaining individual participant's goals with the studied intervention e. Safety of the intervention procedure

Sample size. To determine the required sample size (n) for our study, the research team conducted an a priori estimation based on data from a 2021 paper by Tan et Jia, which was closely aligned with our research. The data were the means difference between groups at 4 weeks post-intervention which indicated a mean difference of -14,56° and a corresponding 95% confidence interval (CI) of 6,70° to 21,41° for our primary endpoint: the improvement in shoulder external rotation passive range of motion, as measured by goniometry.

To calculate the standard deviation (SD), investigators extracted it from the confidence interval using the RevMan tool provided in the Cochrane website (https://training.cochrane.org/resource/revman-calculator), which yielded an SD of 10,857°.

The researchers then used the Sampsize web tool (https://app.sampsize.org.uk/) to calculate the sample size for a non-inferiority parallel trial. A non-inferiority margin of 5°, a power of 0,90, a significance level of 0,05, and an allocation ratio of 1 were considered. This calculation resulted in a required sample size of 23 participants per group.

Baseline Evaluation All participants are evaluated at baseline, 1-2 weeks before the intervention session for the endpoints numbered above using the respective outcome measures.

Arms During the intervention session, participants in the Cryoneurolysis arm undergo ultrasound-guided peripheral nerve cryoneurolysis, while participants in the control arm receive ultrasound-guided intramuscular injections of BoNT-A.

These procedures are explained in detail below and are performed by physicians who have received specialized training in ultrasound-guided cryoneurolysis and BoNT-A intramuscular injections. Specifically, at Rehazenter in Luxembourg, these procedures are carried out by José Pereira, M.D., and Frederic Chantraine, M.D., while in Portugal, Simao Serrano, M.D., and Joao Constantino, M.D., are responsible for performing them. The ultrasound device used is the E10 from General Electric.

Cryoneurolysis The cryoneurolysis intervention is performed by a trained and experienced physician. Ultrasound guided cryoneurolysis to the lateral pectoral nerve and to the thoracodorsal nerve is the intervention in this group. The 3 parts of the pectoral major muscle (clavicular, sternal and costal) innervated by different branches of the lateral pectoral nerve might be targeted as needed.

The cryoneurolysis device being used is the "Cryo-S Painless" produced by Metrum, a manufacturer based in Poland. The cryoprobes have a caliber of 1.3 mm. These devices hold medical certification ( CE) for cryoanalgesia within the European Union.

Technical and certification files are provided to the Regulatory agencies in Luxembourg.

(https://www.metrum.com.pl/produkty/cryo-s-painless-2/?lang=en ). Several precautions steps are taken to prevent the incidence of adverse effects. Motor branches or pure motor nerves will be targeted, since targeting mixed sensory and motor nerves may lead to unwanted numbness or dysesthesia.

The procedure is described in the following steps:

The skin area around the injection site is prepared with a proper aseptic solution, selected according with possible previous participant's allergic reactions. The skin, subcutaneous tissue and muscle planes are anesthetized with a small volume of 1% lidocaine (maximum total dose of 2mg/kg).

The cryoprobe is sterile and before using it in the participant, it is tested by the interventional physician with one cycle of ice ball formation. The ice ball and the probe are checked to any possible unexpected malfunction.

A 14-gauge angiocath is inserted into the anesthetized skin. The cryoprobe is then be passed through the angiocath. This allows to protect the cutaneous tissue from eventual cold induced lesions.

Ultrasound guidance with high a resolution probe is mandatory. It allows to have a live visualization of the procedure, identify the nerves and its sono-anatomy, avoid noble structures as vessels, and screen any underlying structural pathology which precludes the procedure.

Before the cycle of cryoneurolysis, nerve electrical stimulation for muscle and sensory activation adds an extra layer of security, it verifies that the targeted nerve innervates the corresponding spastic muscle(s) and that there is no sensory nerve branch in which cryoneurolysis might induce dysesthesia.

One cycle of cryoneurolysis lasts 120 seconds. Two cycles around the selected nerve are performed with a minimum of 45 seconds interval between cycles corresponding to the thawing phase. The expected theoretical minimal temperature between the tip of the cryoprobe and the interior of the ice ball is around -75°C and the expected temperature of the ice ball neighboring tissue during the cycle is approximately -40°C depending on the heat drain. The employed cryoprobes are single use, straight, 120 mm long, 1,3 mm diameter (18 Ga), with integrated neurostimulation feature (motor and sensory).

After completion of the procedure, the physician waits for the thawing and gently removes the cryoprobe whenever it is easily released from the tissues.

Intramuscular BoNT-A injection Participants allocated to this group have intramuscular injections, guided by ultrasound and electrical neurostimulation, of BoNT-A (ona botulinum toxin A) to the pectoralis major (75 UI), subscapularis (75 UI) and teres major (50 UI), dilution 100UI/ml. These muscles selection and doses are chosen according to a literature review 60,76,77,81 incriminating these 3 muscles as the responsible for a common spastic pattern of shoulder adduction and internal rotation and contributing to the shoulder pain.

The procedure follows the institutional routine practice in terms of BoNT-A intramuscular injection procedure, using ultrasound with or without electrical neuromuscular stimulation and is performed by a trained and experienced medical doctor.

Randomization In order to minimize bias, assignment of participants with eligibility criteria to either group (ultrasound guided / neurostimulation cryoneurolysis or BoNT-A intramuscular injection) is randomized. The process of randomization is managed by an independent member of the research team, blinded, and not related to intervention sessions or outcome measures assessment. To avoid selection bias, a clinical trial randomization webtool is used so no human will have any interference in the subject's trial arm allocation.

The process of randomization will be based in block allocation of 4, with stratification to level of impairment. This strategy allows, as the trial is ongoing, to balance the two groups in terms of number of patients and patients' impairment profile. In the stratification for impairment level, participants will be hierarchically classified in 4 clusters according to the Fugl-Meyer score from baseline assessment: severe (0-15), severe-moderate (16-34) ; moderate-mild (35-53); mild (54-66).

Masking By the nature of this study, blinding either participants or outcome measures evaluators is not realistic and so there is no masking. Blinding the interventionist physician is impossible for obvious reasons. Since participants in the two groups have an intervention that aims a therapeutic effect, a placebo/nocebo effect bias is not expected. For this reason, investigators acknowledge potential limitations, such as potential bias in outcome measurements due to the lack of masking.

Comprehensive Evaluation The comprehensive evaluation at both baseline and throughout the trial is conducted by the same evaluators who will be limited to three individuals. These evaluators are highly trained in deploying the outcome measures and are part of the institutional staff, comprising physiotherapists and occupational therapists. The evaluations will take place at dedicated stations, following the timeline outlined in the study flowchart and will be documented electronically. The Case Report Form (CRF) document details comprehensive assessment of the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old.
* Have a clinically and functionally stable condition.
* Present spastic hemiplegia of the upper limb caused by a stroke, traumatic, or hypoxic brain event occurring more than 6 months before the study.
* The paretic upper limb must present significant spastic plegia at the shoulder adductors and/or shoulder internal rotators (≥ 1+ on the Modified Ashworth Scale).
* Have a Visual Analogue Scale (VAS) pain score > 40/100 mm.
* Have spasticity causing limitations in providing care.
* Have the cognitive capacity to make informed decisions. A comprehensive explanation of the study will be provided orally and in writing to participants and a trusted relative of their choosing.
* Maintain any medications on a stable schedule.
* Accept and have access to an interdisciplinary rehabilitation program and standardized evaluation sessions throughout the study.

Exclusion Criteria:

* In the investigator's opinion, the subject will be exposed to unacceptable risk by participation.
* Previous intervention or condition that altered the target neural anatomy of the upper limb.
* Any injection (neurolytic, sclerosing, anesthesia, etc.) to the upper limb within the last 4 months.
* Spasticity invasive treatment such as intrathecal baclofen during the trial.
* Current enrollment in an investigational drug or device study targeting spasticity management.
* Pregnancy or lactation.
* Allergy or intolerance to local anesthesia/BoNT-A.
* Contraindications to BoNT-A administration, such as:

  * Myasthenia Gravis
  * Eaton-Lambert syndrome
  * Possible drug interactions (e.g., aminoglycosides and BoNT-A)
* Any local skin condition at the treatment site that may adversely affect treatment or outcomes.
* Chronic medication use (prescription or over-the-counter) that, in the investigator's opinion, would affect study participation or subject safety.
* Contraindications to cryoneurolysis, including:

  * Diagnosis of cryoglobulinemia
  * Paroxysmal cold hemoglobinuria
  * Cold urticaria
  * Raynaud's disease
  * Any form of peripheral neuropathy
  * Open and/or infected wounds on the affected limb
* Diagnosis of concomitant progressive neurological diseases such as Amyotrophic Lateral Sclerosis.
* Any reason, in the investigator's opinion, that the subject may not be suitable for study participation (e.g., history of noncompliance, drug addiction, or any related upper limb injury).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Change in active Range of motion shoulder | baseline, week 1, 4, 12 and 24
  Active Range of Motion (AROM) measure in angles (Deg) at the shoulder assesses joint mobility through voluntary movement by the patient. The healthcare professional instructs the patient to perform the following motions:
  Flexion: Arm moves forward and upward. Extension: Arm moves backward. Abduction: Arm lifts outward to the side. Adduction: Arm moves across the body. Internal Rotation: Arm rotates inward (e.g., hand behind back). External Rotation: Arm rotates outward (e.g., hand behind head). The clinician observes for range, quality, symmetry, and compensatory movements. A goniometer measures the motion in degrees, compared to normative or baseline values. AROM helps identify muscle strength, joint limitations, and functional deficits, providing a reliable outcome measure in rehabilitation.
Change in passive range of motion of shoulder | baseline, week 1,4,12,24
  Passive Range of Motion (PROM), measured in angles (Deg) performed by a healthcare professional, assesses joint mobility in the shoulder.
  The clinician gently moves the shoulder through its full range while the patient remains relaxed, measuring:
  Flexion (forward arm movement) Extension (backward arm movement) Abduction (arm movement away from the body) Adduction (arm movement toward the body) Internal rotation (arm rotates inward) External rotation (arm rotates outward). A goniometer records the motion in degrees, compared to normative values or baseline measurements. PROM is essential for identifying joint stiffness, contractures, or spasticity and tracking mobility changes over time, making it a reliable outcome measure in rehabilitation.

SECONDARY OUTCOMES:
Change in muscle tone muscles controlling the shoulder | Baseline, week 1, 4, 12, 24
  Modified Ashworth scale, number in a scale from 0 to 4. score: 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement) 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Change in nociceptive pain: Visual analogue scale | Baseline, week 1,4,12,24
  The Visual Analog Scale (VAS) measured in mm in a 100 mm bar, is a simple, widely used tool for assessing nociceptive pain intensity. Since you are using a vertical bar with the maximum pain at the top, the scale will appear as a straight vertical line, typically 10 centimeters long. It is anchored by two descriptors:
  At the bottom: "No Pain" At the top: "Worst Imaginable Pain" Patients are instructed to mark a point on the vertical line that corresponds to the intensity of their current pain. This mark reflects their subjective experience of pain at that moment. To quantify the pain level, measure the distance from the bottom of the line to the patient's mark, usually in centimeters or millimeters. This measurement provides a numerical value of pain intensity on a scale from 0 to 10.
Upper limb fonction - Fugl-Meyer Assessment (FMA) | Baseline, Week 24
  The Fugl-Meyer Assessment (FMA) measured in numbers in a scale 0-66. Upper Limb part is a standardized tool to measure changes in upper limb function after stroke or neurological injury. It evaluates motor recovery across shoulder, elbow, wrist, and hand movements.
  Components:
  Volitional Movement: Assess active motions (e.g., flexion, extension, abduction, and rotation) of the upper limb.
  Coordination/Speed: Perform finger-to-nose or repetitive tasks. Reflex Activity: Evaluate reflex presence at specific joints.
  Each item is scored on a 3-point scale:
  0: Cannot perform.
  1. Partial movement.
  2. Full movement. The maximum score for the upper limb is 66 points. Higher scores indicate better motor function. The FMA is sensitive to functional changes over time, making it a reliable outcome measure in rehabilitation.
Quality of Life | Baseline, Week 24
  The SF-36 (Short Form-36) is a standardized questionnaire used to measure changes in quality of life across 8 domains:
  Physical Functioning Role Limitations (Physical) Bodily Pain General Health Vitality Social Functioning Role Limitations (Emotional) Mental Health Patients rate their experiences over the past 4 weeks using Likert scales or yes/no responses. Scores for each domain are transformed into a 0-100 scale, with higher scores indicating better quality of life.
  The SF-36 provides a physical component summary (PCS) and a mental component summary (MCS), allowing for comprehensive evaluation of changes in overall health. It is widely used in clinical and research settings for tracking improvements or declines over time.
Tardieu Modified scale | baseline, week 1, 4, 12 and 24
  1. Quality of muscle reaction
  2. Angle of muscle reaction 3 speed definitions:
  1) V1 is slow as possible 2) V2 speed of limb falling under gravity 3) V3 moving as fast as possible Quality of Muscle Reaction (scored 0-5); 0 is no resistance to passive ROM to 5 indicating joint is immobile (Some versions scored 0-4).
  Grade 0: No resistance throughout the course of the passive movement Grade 1: Slight resistance throughout the course of the passive movement, followed by release Grade 2: Clear catch at precise angle, interrupting the passive movement, followed by release Grade 3: Fatigable clonus (< 10 seconds when maintaining pressure) occurring at precise angle Grade 4: Infatigable clonus (> 10 seconds when maintaining pressure occurring at precise angle Joint Angle: Modified Tardieu describes R1 and R2; R1 is the angle of muscle reaction, R2 is the full PROM.
  The angle of full ROM (R2) is
Change in neuropathic pain - Douleur Neuropathique 4 (DN4) | baseline, week 1, 4, 12 and 24
  he DN4 (Douleur Neuropathique 4) is a rapid and validated questionnaire used to assess neuropathic pain. It consists of 10 items:
  7 sensory descriptors (burning, painful cold, electric shocks, tingling, pins and needles, numbness, itching), based on the patient's history.
  3 clinical examination findings (hypoesthesia to touch, hypoesthesia to pinprick, and allodynia).
  Each positive answer scores 1 point. A total score ≥4/10 indicates a high likelihood of neuropathic pain. The DN4 is easy to administer, taking only 2-3 minutes, and provides a quick differential tool for distinguishing neuropathic pain from nociceptive pain in clinical practice. It is widely used in both research and routine care.
Change in upper limb function - Box and Block Test | Baseline, Week 24
  The Box and Block Test (BBT) is a standardized tool to measure gross manual dexterity in the upper limb. Measured in number of blocks being moved correctly.
  Procedure:
  The patient is seated at a table with a partitioned box containing 150 small blocks (2.5 cm³).
  Using one hand, the patient moves as many blocks as possible from one side of the box to the other within 60 seconds.
  The test is performed separately for each hand.
  Scoring:
  The number of blocks successfully transferred is counted. Higher scores indicate better manual dexterity.
  The BBT is quick, reliable, and sensitive to changes in function over time, making it an effective outcome measure for assessing upper limb performance in rehabilitation, particularly for conditions like stroke or neurological impairments.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehazenter, Centre National de Rééducation fonctionnelle et de Réadaptation, Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: Yes
All the outcome measures data will be shared
Supporting Information: Study Protocol, ICF
Time Frame: Shared after post-hoc analysis data

REFERENCES:
- [Background] Verduzco-Gutierrez M, Raghavan P, Pruente J, Moon D, List CM, Hornyak JE, Gul F, Deshpande S, Biffl S, Al Lawati Z, Alfaro A. AAPM&R consensus guidance on spasticity assessment and management. PM R. 2024 Aug;16(8):864-887. doi: 10.1002/pmrj.13211. Epub 2024 May 21. PMID 38770827